CLINICAL TRIAL: NCT01424514
Title: A Randomised, Double Blind Placebo Controlled, 2 Way Cross Over Study in Adults With Non-allergic Rhinits to Evaluate the Effect of Once Daily Administration of Intranasal SB-705498 12mg for Two Weeks and the Response to a Chamber Challenge of Cold Dry Air
Brief Title: SB705498 Proof of Concept Chamber Challenge in Subjects With Non Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 114974
Record Dates: First submitted 2011-08-18; First posted 2011-08-29 (Estimated); Results first posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2017-04

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis | interventions — SB 705498

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SB-705498 (Experimental)
  Interventions: Drug: SB-705498
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SB-705498 — 12mg intra nasal
  Arms: SB-705498
Drug: Placebo — Placebo intra nasal
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the pharmacodynamic (PD) effects (Total Symptom Score (TSS) and its individual components: rhinorrhoea, nasal congestion, post-nasal drip) of intranasal, repeat dose SB-705498 in non-allergic rhinitis (NAR) patients elicited by a cold dry air challenge in an environmental exposure chamber (EEC). SB-705498 is a selective antagonist of the transient receptor potential vanilloid-1 (TRPV1) ligand gated ion channel. TRPV1 is a cation permeable ion channel that can be activated by several physiological factors, such as heat, protons (pH), osmotic stress, eicosanoid derivatives, anandamide, and by products of inflammation, such as histamine, prostaglandins and bradykinin. In the nose, the local TRPV1 expressing sensory C-fibres are thought to play a key role in the development of nasal hyper-responsiveness to environmental provocateurs. It has been proposed that blocking the nasal sensory nerve stimulation may control nasal hyper-responsiveness and therefore prevent the induction of rhinitis symptoms. In this context, preclinical evidence supports that targeting TRPV1 by SB-705498 may be an attractive option.

In this study NAR patients will be randomised, in a double blind, placebo controlled cross over design to receive 14 day repeat doses of 12mg intra-nasal SB-705498 once daily. Whilst dosing at home, subjects will record symptom scores to document their symptoms. In addition, during visits to the clinical unit, acoustic rhinometry, quality of life questionnaires and safety assessments will be monitored.

ELIGIBILITY:
Inclusion Criteria:

Deviations from inclusion criteria are not allowed because they can potentially jeopardize the scientific integrity of the study, regulatory acceptability or subject safety. Therefore, adherence to the criteria as specified in the protocol is essential.

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Diagnosis of NAR, as determined by the presence of perennial rhinitis symptoms that last for several months per year, for more than 1 year and are not attributed to allergy, infections or nasal abnormalities. Positive history of rhinitis symptoms triggered by environmental provocateurs (e.g. weather changes, irritants, air pollution etc), but not allergens.
2. Normal levels of total plasma IgE and negative allergy skin or Rast tests to common aeroallergens.
3. Male or female between 18 and 65 years of age inclusive.
4. A female subject is eligible to participate if she is of:

   * Non-childbearing potential defined as pre-menopausal females with a \documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
   * Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 84 days post-last treatment administration.
5. Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 84 days post-last treatment administration.
6. Body weight ≥ 50 kg (males) and ≥45kg (females) and BMI within the range 19 - 29.9 kg/m2 (inclusive).
7. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
8. Available to complete all the required study measurements.
9. Single QTc, < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
10. The subject must demonstrate at screening TSS ≥ 4 (on a 9 point scale) at screening visits 1 and 2.
11. AST and ALT < 2xULN; alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

Deviations from exclusion criteria are not allowed because they can potentially jeopardise the scientific integrity of the study, regulatory acceptability or subject safety. Therefore, adherence to the criteria as specified in the protocol is essential.

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Nasal abnormalities likely to affect the outcome of the study, i.e. nasal septal perforation, nasal polyps, other nasal malformations.
2. History of frequent nosebleeds.
3. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
4. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
5. Positive pre-study drug/alcohol/smoking screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids, benzodiazepines and methadone
6. A positive test for HIV antibody.
7. History of regular alcohol consumption within 6 months of the study defined as:

   • An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
8. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
9. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
10. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.

    Subjects who are using some of the medications below on an as needed basis, may participate in the study if they remain free of medication for the following periods of time prior to each visit:
    * Nasal antihistamines: 48 hours
    * Oral antihistamines A (cetirizine, fexofenadine, loratadine, desloratadine): 7 days
    * Oral antihistamines B (all others): 7 days
    * Nasal decongestants: 24 hours
    * Oral decongestants: 24 hours
    * Nasal glucocorticosteroids: 4 weeks
    * Inhaled glucocorticoids: 4 weeks
    * Oral glucocorticosteroids: 12 weeks
    * Oral leukotriene receptor antagonists: 7 days
    * Oral 5-lipoxygenase inhibitors: 7 days
    * Oral methylxanthines: 7 days Subjects with recent upper respiratory tract infections (URTIs) will be allowed in the study only if their nasal symptoms have been completely resolved for more than 3 weeks prior to screening.
11. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
12. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
13. Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
14. Lactating females.
15. Unwillingness or inability to follow the procedures outlined in the protocol.
16. Subject is mentally or legally incapacitated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-12-01; Primary Completion 2011-04-01 (Actual); Study Completion 2011-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 114974 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114974 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114974 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114974 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114974 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114974 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114974 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned on 40 participants, male or female between 18 and 65 years of age with non-allergic rhinitis (NAR), at a single center of Canada from 7th December 2010 to 18th April 2011.
Groups:
- Active Then Placebo: Participants received repeat doses of intranasal spray of SB-705498 12 milligram (mg) as an active intervention once daily for 14 days during intervention period 1 according to a plan of randomization. After a washout period of 4 weeks, participants then received repeat doses of matching placebo once daily for 14 days during intervention period 2.
- Placebo Then Active: Participants received repeat doses of matching placebo once daily for 14 days during intervention period 1 according to a plan of randomization. After a washout period of 4 weeks, participants then received repeat doses of intranasal spray of SB-705498 12 mg as an active intervention once daily for 14 days during intervention
Period: Period 1:Intervention Period 1 (14 Days)
Arm/Group | Active Then Placebo | Placebo Then Active
Started | 20 | 20
Completed | 19 | 19
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1
Period: Period 2:Washout Period (4 Weeks)
Arm/Group | Active Then Placebo | Placebo Then Active
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Period 3:Intervention Period 2 (14 Days)
Arm/Group | Active Then Placebo | Placebo Then Active
Started | 19 | 19
Completed | 18 | 19
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Treatments Combined: The study consisted of 2 treatment periods, each of 14 days (2 weeks). The treatment periods were separated by at least 4 weeks of washout period. Participants were administered intranasal spray of SB-705498 12 milligram (mg) or matching placebo as repeat doses for 14 days once daily in treatment period 1 (TP1), and the converse treatments in TP2 two treatment sequences (active/placebo [A/P] or placebo/active [P/A]) with respect to the randomization.
Arm/Group | All Treatments Combined
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.6 (11.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 3
  American Indian or Alaska Native | 1
  Asian - Central/South Asian Heritage | 1
  Asian - East Asian Heritage | 2
  Asian - South East Asian Heritage | 1
  White - Arabic/North African Heritage | 2
  White - White/Caucasian/European Heritage | 29
  Mixed Race | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Total Symptom Score (TSS) Elicited by a 1 Hour (h) Cold Dry Air (CDA) Challenge, 1 h and 24 h on Day 14 to Compare the Effect of 14 Day Repeat Dosing of Intranasal SB-705498 12 mg With Placebo
Description: TSS was calculated based on a CDA challenge, done for 1 h in a controlled environmental exposure chamber which was validated for 14+/-5 degree Celsius (C), <15% relative humidity and 5+/-3 feet per second (ft/sec) air velocity, 1 h and 24 h post dose on Day 14 (Day 15). TSS was calculated as the sum of the response for 3 components of nasal congestion, rhinorrhoea and post nasal drip. It was rated on a 4-point scale ranging from 0 to 3, where: 0=absent, 1=mild, 2=moderate, and 3=severe (symptom hard to tolerate). TSS score ranges from 0-9 with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms. Weighted mean (WM) for TSS was calculated over the time interval 0 to 60 minute (m) after start of CDA challenge by calculating area under the curve (AUC) of the TSS via the linear trapezoidal method then dividing by the total duration that the participant took to complete CDA challenge assessments. WM is reported as least square (LS) mean.
Time Frame: Day 14 to Day 15 of each period (Day 14, 24 h post- dose was done on Day 15)
Population: All Subjects population defined as all participants who received at least one dose of study medication. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Groups:
- Placebo: Eligible participants received matching placebo to SB-705498 12 mg once daily for 14 days in each of the 2 treatment periods, where participants were randomized to any of the two treatment sequences (active/placebo or placebo/active) separated by at least 4 weeks of washout period.
- SB-705498 12 mg: Eligible participants received intranasal spray of SB-705498 12 mg once daily for 14 days in each of the 2 treatment periods, where participants were randomized to any of the two treatment sequences (active/placebo or placebo/active) separated by at least 4 weeks of washout period.
Arm/Group | Placebo | SB-705498 12 mg
Number analyzed (Participants) | 38 | 39
Scores on scale
  WM 0-60 TSS, 1 h: number analyzed (Participants) | 37 | 39
  WM 0-60 TSS, 1 h | 3.49 (0.259) | 3.37 (0.254)
  WM 0-60 TSS, 24 h: number analyzed (Participants) | 38 | 38
  WM 0-60 TSS, 24 h | 3.56 (0.263) | 3.59 (0.262)
  Maximum TSS, 1 h: number analyzed (Participants) | 37 | 39
  Maximum TSS, 1 h | 4.55 (0.285) | 4.51 (0.279)
  Maximum TSS, 24 h: number analyzed (Participants) | 38 | 38
  Maximum TSS, 24 h | 4.71 (0.295) | 4.82 (0.295)
Statistical Analysis 1: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for 1 h in WM 0-60 TSS; Test type: Superiority or Other; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.60 to 0.36], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for 24 h in WM 0-60 TSS; Test type: Superiority or Other; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.45 to 0.51], Standard Error of Mean 0.24
Statistical Analysis 3: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for 1 h in Maximum TSS; Test type: Superiority or Other; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.58 to 0.51], Standard Error of Mean 0.27
Statistical Analysis 4: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for 24 h in Maximum TSS; Test type: Superiority or Other; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.51 to 0.72], Standard Error of Mean 0.30

2. Primary Outcome: Mean Individual Component of TSS of Rhinorrhoea (Runny Nose), Nasal Congestion and Post-nasal Drip Elicited by a 1 h CDA Challenge, 1 h and 24 h on Day 14 to Compare the Effect of 14 Day Repeat Dosing of Intranasal SB-705498 12 mg With Placebo
Description: The individual components of TSS was calculated based on a CDA challenge, done for 1 h in a controlled environmental exposure chamber which was validated for 14+/-5 degree C, <15% relative humidity and 5+/-3 ft/sec air velocity, 1 h and 24 h post dose on Day 14 (Day 15). The individual component of TSS nasal symptoms were nasal congestion, rhinorrhoea (runny nose), and post nasal drip It was rated on a 4-point scale ranging from 0 to 3, where: 0=absent, 1=mild, 2=moderate, and 3=severe (symptom hard to tolerate). The scores of the individual components of TSS ranges from 0-3 with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms. WM for TSS was calculated over the time interval 0 to 60 m after start of CDA challenge by calculating AUC of the TSS via the linear trapezoidal method then dividing by the total duration that the participant took to complete CDA challenge assessments. WM is reported as LS mean.
Time Frame: Day 14 to Day 15 of each period (Day 14, 24 h post- dose was done on Day 15)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | SB-705498 12 mg
Number analyzed (Participants) | 38 | 39
Score on scale
  WM 0-60 nasal congestion, 1 h: number analyzed (Participants) | 37 | 39
  WM 0-60 nasal congestion, 1 h | 1.09 (0.667) | 1.08 (0.744)
  WM 0-60 nasal congestion, 24 h: number analyzed (Participants) | 38 | 38
  WM 0-60 nasal congestion, 24 h | 1.24 (0.708) | 1.18 (0.691)
  Maximum nasal congestion, 1 h: number analyzed (Participants) | 37 | 39
  Maximum nasal congestion, 1 h | 1.46 (0.836) | 1.33 (0.838)
  Maximum nasal congestion, 24 h: number analyzed (Participants) | 38 | 38
  Maximum nasal congestion, 24 h | 1.61 (0.823) | 1.53 (0.862)
  WM 0-60 runny nose, 1 h: number analyzed (Participants) | 37 | 39
  WM 0-60 runny nose, 1 h | 1.24 (0.600) | 1.19 (0.600)
  WM 0-60 runny nose, 24 h: number analyzed (Participants) | 38 | 38
  WM 0-60 runny nose, 24 h | 1.19 (0.596) | 1.29 (0.616)
  Maximum runny nose, 1 h: number analyzed (Participants) | 37 | 39
  Maximum runny nose, 1 h | 1.68 (0.709) | 1.77 (0.583)
  Maximum runny nose, 24 h: number analyzed (Participants) | 38 | 38
  Maximum runny nose, 24 h | 1.76 (0.634) | 1.95 (0.655)
  WM 0-60 post nasal drip, 1 h: number analyzed (Participants) | 37 | 39
  WM 0-60 post nasal drip, 1 h | 1.14 (0.642) | 1.06 (0.721)
  WM 0-60 post nasal drip, 24 h: number analyzed (Participants) | 38 | 38
  WM 0-60 post nasal drip, 24 h | 1.07 (0.637) | 1.10 (0.803)
  Maximum post nasal drip, 1 h: number analyzed (Participants) | 37 | 39
  Maximum post nasal drip, 1 h | 1.51 (0.692) | 1.44 (0.882)
  Maximum post nasal drip, 24 h: number analyzed (Participants) | 38 | 38
  Maximum post nasal drip, 24 h | 1.45 (0.724) | 1.47 (0.862)

3. Secondary Outcome: Mean Total Symptom Score (TSS) Elicited by a 1 Hour (h) CDA Challenge, 1 h Post-dose on Day 1 to Compare the Effect of a Single Dose of 12 mg Intranasal SB-705498 With Placebo
Description: TSS was calculated based on a CDA challenge, done for 1 h in a controlled environmental exposure chamber which was validated for 14+/-5 degree C, <15% relative humidity and 5+/-3 ft/sec air velocity, 1 h and 24 h post dose on Day 1. TSS was calculated as the sum of the response for 3 components of nasal congestion, rhinorrhoea and post nasal drip. It was rated on a 4-point scale ranging from 0 to 3, where: 0=absent, 1=mild, 2=moderate, and 3=severe (symptom hard to tolerate). TSS score ranges from 0-9 with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms. WM for TSS was calculated over the time interval 0 to 60 m after start of CDA challenge by calculating AUC of the TSS via the linear trapezoidal method then dividing by the total duration that the participant took to complete CDA challenge assessments. WM is reported as LS mean.
Time Frame: Day 1 of each period
Population: All Subjects Population.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Placebo | SB-705498 12 mg
Number analyzed (Participants) | 38 | 40
Scores on scale
  WM 0-60 TSS | 3.44 (0.229) | 3.56 (0.227)
  Maximum TSS | 4.80 (0.252) | 4.89 (0.249)
Statistical Analysis 1: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for WM 0-60 TSS; Test type: Superiority or Other; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.30 to 0.54], Standard Error of Mean 0.21
Statistical Analysis 2: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for Maximum TSS; Test type: Superiority or Other; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.39 to 0.57], Standard Error of Mean 0.24

4. Secondary Outcome: Mean Individual Component of TSS of Rhinorrhoea (Runny Nose), Nasal Congestion and Post-nasal Drip Elicited by a 1 h CDA Challenge, 1 h Post-dose on Day 1 to Compare the Effect of a Single Dose of 12 mg Intranasal SB-705498 With Placebo
Description: The individual components of TSS was calculated based on a CDA challenge, done for 1 h in a controlled environmental exposure chamber which was validated for 14+/-5 degree C, <15% relative humidity and 5+/-3 ft/sec air velocity, 1 h and 24 h post dose on Day 1. The individual component of TSS nasal symptoms were nasal congestion, rhinorrhoea (runny nose), and post nasal drip It was rated on a 4-point scale ranging from 0 to 3, where: 0=absent, 1=mild, 2=moderate, and 3=severe (symptom hard to tolerate). The score ranges from 0-3 with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms. WM for TSS was calculated over the time interval 0 to 60 m after start of CDA challenge by calculating AUC of the TSS via the linear trapezoidal method then dividing by the total duration that the participant took to complete CDA challenge assessments. WM is reported as LS mean.
Time Frame: Day 1 of each period
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo | SB-705498 12 mg
Number analyzed (Participants) | 38 | 39
Scores on scale
  WM 0-60 nasal congestion | 1.09 (0.687) | 1.10 (0.562)
  Maximum nasal congestion | 1.47 (0.830) | 1.51 (0.756)
  WM 0-60 runny nose | 1.21 (0.609) | 1.34 (0.451)
  Maximum runny nose | 1.89 (0.689) | 1.91 (0.427)
  WM 0-60 post nasal drip | 1.11 (0.665) | 1.10 (0.583)
  Maximum post nasal drip | 1.53 (0.797) | 1.55 (0.677)

5. Secondary Outcome: Mean TSS From Day 7 to Day 14 (Post-dose Prior to Challenge) Following Repeat Doses of SB-705498
Description: TSS was calculated as the sum of the response for 3 components of nasal congestion, rhinorrhoea and post nasal drip. It was rated on a 4-point scale ranging from 0 to 3, where: 0=absent, 1=mild, 2=moderate, and 3=severe (symptom hard to tolerate). TSS score ranges from 0-9 with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms. For Day 1 to 14 of each study period, participants were asked to keep a diary to record their symptoms whilst at home provided by the clinical unit. Reflective rating represented the symptoms over the proceeding 12 h which was performed once daily in the evening (PM). The PM reflective rating was done approximately 12 h after dosing, but before bedtime. If any of the individual components were missing then the TSS was set to be missing for that participant at that timepoint.
Time Frame: Day 7 to Day 14 of each period
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo | SB-705498 12 mg
Number analyzed (Participants) | 38 | 39
Scores on scale
  Day 1 | 1.4 (1.53) | 1.2 (1.29)
  Day 7 | 3.3 (1.86) | 3.4 (1.83)
  Day 8 | 3.1 (1.87) | 3.3 (1.99)
  Day 9 | 2.9 (1.50) | 3.5 (2.01)
  Day 10 | 3.1 (1.87) | 3.2 (1.93)
  Day 11: number analyzed (Participants) | 38 | 38
  Day 11 | 3.1 (2.14) | 3.0 (2.01)
  Day 12: number analyzed (Participants) | 38 | 38
  Day 12 | 3.6 (2.02) | 2.9 (1.83)
  Day 13 | 3.3 (2.01) | 2.9 (1.97)
  Day 14: number analyzed (Participants) | 37 | 39
  Day 14 | 2.0 (1.88) | 1.8 (1.82)

6. Secondary Outcome: Mean Individual Component of TSS of Rhinorrhoea (Runny Nose), Nasal Congestion and Post-nasal Drip From Day 7 to Day 14 Following Repeat Doses of SB-705498
Description: The individual component of TSS nasal symptoms of nasal congestion, rhinorrhoea (runny nose) and post nasal drip was scored on a 4-point scale ranging from 0 to 3, where: 0=absent, 1=mild, 2=moderate, and 3=severe (symptom hard to tolerate). The scores of the individual components of TSS ranges from 0-3 with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms. For Day 1 to 14 of each study period, participants were asked to keep a diary to record their symptoms whilst at home on a diary card provided by the clinical unit. Reflective rating represented the symptoms over the proceeding 12 h which was performed once daily in the PM. The PM reflective rating was done approximately 12 h after dosing, but before bedtime.
Time Frame: Day 7 to Day 14 of each period
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo | SB-705498 12 mg
Number analyzed (Participants) | 38 | 39
Scores on scale
  Nasal congestion, Day 1 | 0.6 (0.72) | 0.5 (0.60)
  Nasal congestion, Day 7 | 1.2 (0.79) | 1.2 (0.78)
  Nasal congestion, Day 8 | 1.1 (0.84) | 1.2 (0.78)
  Nasal congestion, Day 9 | 0.9 (0.61) | 1.2 (0.78)
  Nasal congestion, Day 10 | 1.1 (0.73) | 1.2 (0.88)
  Nasal congestion, Day 11: number analyzed (Participants) | 38 | 38
  Nasal congestion, Day 11 | 1.1 (0.81) | 1.1 (0.87)
  Nasal congestion, Day 12: number analyzed (Participants) | 38 | 38
  Nasal congestion, Day 12 | 1.2 (0.75) | 1.2 (0.75)
  Nasal congestion, Day 13 | 1.2 (0.75) | 1.1 (0.81)
  Nasal congestion, Day 14: number analyzed (Participants) | 37 | 39
  Nasal congestion, Day 14 | 0.8 (0.90) | 0.8 (0.82)
  Runny nose, Day 1 | 0.3 (0.52) | 0.3 (0.50)
  Runny nose, Day 7 | 1.1 (0.83) | 1.2 (0.80)
  Runny nose, Day 8 | 1.1 (0.76) | 1.1 (0.80)
  Runny nose, Day 9 | 1.1 (0.70) | 1.2 (0.84)
  Runny nose, Day 10, | 1.1 (0.78) | 1.1 (0.75)
  Runny nose, Day 11,: number analyzed (Participants) | 38 | 38
  Runny nose, Day 11, | 1.1 (0.91) | 1.1 (0.78)
  Runny nose, Day 12,: number analyzed (Participants) | 38 | 38
  Runny nose, Day 12, | 1.2 (0.83) | 1.0 (0.77)
  Runny nose, Day 13, | 1.1 (0.89) | 1.1 (0.85)
  Runny nose, Day 14,: number analyzed (Participants) | 37 | 39
  Runny nose, Day 14, | 0.6 (0.73) | 0.3 (0.62)
  Post nasal drip, Day 1 | 0.5 (0.65) | 0.4 (0.60)
  Post nasal drip, Day 7 | 0.9 (0.82) | 1.0 (0.84)
  Post nasal drip, Day 8 | 0.8 (0.77) | 1.0 (0.83)
  Post nasal drip, Day 9 | 0.9 (0.76) | 1.1 (0.92)
  Post nasal drip, Day 10 | 0.9 (0.75) | 0.9 (0.83)
  Post nasal drip, Day 11: number analyzed (Participants) | 38 | 38
  Post nasal drip, Day 11 | 0.9 (0.83) | 0.8 (0.82)
  Post nasal drip, Day 12: number analyzed (Participants) | 38 | 38
  Post nasal drip, Day 12 | 1.1 (0.91) | 0.8 (0.78)
  Post nasal drip, Day 13 | 1.0 (0.84) | 0.8 (0.81)
  Post nasal drip, Day 14: number analyzed (Participants) | 37 | 39
  Post nasal drip, Day 14 | 0.6 (0.73) | 0.7 (0.77)

7. Secondary Outcome: Mean Sneezing Elicited by a 1 h CDA Challenge at 1 h Post-dose on Day 1, 1 and 24 h Post-dose on Day 14 to Compare the Effect of Intranasal SB-705498 12 mg With Placebo
Description: The assessment of sneezing was done based on a CDA challenge, for 1 h in a controlled environmental exposure chamber which was validated for 14+/-5 degree C, <15% relative humidity and 5+/-3 ft/sec air velocity, 1 h post dose on Day 1 and 1 h and 24 h post dose on Day 14 (Day 15). Sneezing was scored on a 4-point scale ranging from 0 to 3, where: 0=absent, 1=mild, 2=moderate, and 3=severe (symptom hard to tolerate). The score ranges from 0-3 with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms. It was used to derive the WM CDA challenge value calculated over the time interval 0 to 60 m after start of CDA challenge and the maximum score. WM is reported as LS mean.
Time Frame: Day 1, Day 14 and Day 15 of each period (Day 14, 24 h post- dose was done on Day 15)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Placebo | SB-705498 12 mg
Number analyzed (Participants) | 38 | 40
Scores on scale
  WM 0-60, Day 1, 1 h | 0.28 (0.090) | 0.25 (0.090)
  WM 0-60, Day 14, 1 h: number analyzed (Participants) | 37 | 39
  WM 0-60, Day 14, 1 h | 0.23 (0.085) | 0.21 (0.084)
  WM 0-60, Day 14, 24 h: number analyzed (Participants) | 38 | 38
  WM 0-60, Day 14, 24 h | 0.28 (0.083) | 0.23 (0.083)
  Maximum, Day 1, 1 h | 0.50 (0.131) | 0.43 (0.130)
  Maximum, Day 14, 1 h: number analyzed (Participants) | 37 | 39
  Maximum, Day 14, 1 h | 0.35 (0.123) | 0.34 (0.122)
  Maximum, Day 14, 24 h: number analyzed (Participants) | 38 | 38
  Maximum, Day 14, 24 h | 0.45 (0.111) | 0.43 (0.111)
Statistical Analysis 1: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for Day 1, 1 h in WM 0-60 sneezing; Test type: Superiority or Other; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.14 to 0.08], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for Day 14, 1 h in WM 0-60 sneezing; Test type: Superiority or Other; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.13 to 0.09], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for Day 14, 24 h in WM 0-60 sneezing; Test type: Superiority or Other; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.20 to 0.11], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for Day 1, 1 h in Maximum sneezing; Test type: Superiority or Other; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.28 to 0.14], Standard Error of Mean 0.10
Statistical Analysis 5: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for Day 14, 1 h in Maximum sneezing; Test type: Superiority or Other; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.15 to 0.13], Standard Error of Mean 0.07
Statistical Analysis 6: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for Day 1, 24 h in Maximum sneezing; Test type: Superiority or Other; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.20 to 0.16], Standard Error of Mean 0.09

8. Secondary Outcome: Mean Change From Baseline to Day 14 of Acoustic Rhinometry (AR) Following Repeat Dosing of SB-705498 at 2 h and 25 h Post-dose
Description: Overall AR score was obtained by adding minimal cross-sectional area (MCA) for right and left nostril. MCA1 was captured within the nose at a distance of 0 and 2.2 cm and MCA2 at 2.2 and 5.5 cm. MCA1 and MCA2 were captured simultaneously for each nostril, 3 measurements were obtained from each nostril which resulted in 12 data points. Absolute MCA for all regions in left or right nostril was calculated using the 3 acceptable measurements, calculating average of each of right and left MCA's and also by selecting minimum value from these averages to obtain minimum MCA for left and right nostril. Baseline is defined as the value on Day 1 pre- dose. Change from baseline was calculated by subtracting the baseline (Day 1 pre-dose) values from individual post-randomization values done immediately following CDA challenge. In case of missing baseline or post randomization value, the change from baseline was set to be missing. Adjusted mean is reported as LS mean.
Time Frame: Baseline (Day 1 pre-dose), Day 14 and Day 15 of each period (Day 14, 25 h post dose on Day 14 was evaluated on Day 15)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Centimetre square (cm^2)
Groups:
- Placebo: Eligible participants received matching placebo to SB-705498 12 mg once daily for 14 days in each of the 2 treatment periods, where participants were randomized to any of the two treatment sequences (active/placebo or placebo/active)separated by at least 4 weeks of washout period.
Arm/Group | Placebo | SB-705498 12 mg
Number analyzed (Participants) | 38 | 40
Centimetre square (cm^2)
  Day 1, 2 h | 0.01 (0.021) | 0.03 (0.020)
  Day 14, 2 h: number analyzed (Participants) | 37 | 39
  Day 14, 2 h | 0.09 (0.021) | 0.02 (0.021)
  Day 14, 25 h: number analyzed (Participants) | 36 | 38
  Day 14, 25 h | 0.03 (0.022) | 0.05 (0.022)
Statistical Analysis 1: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for Day 1, 2 h in AR; Test type: Superiority or Other; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.03 to 0.07], Standard Error of Mean 0.026
Statistical Analysis 2: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for Day 14, 2 h in AR; Test type: Superiority or Other; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.13 to -0.02], Standard Error of Mean 0.027
Statistical Analysis 3: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for Day 14, 25 h in AR; Test type: Superiority or Other; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.04 to 0.08], Standard Error of Mean 0.031

9. Secondary Outcome: Mean Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Following Repeat Doses of SB-705498 on Day 14
Description: The RQLQ is a 28-item, disease-specific quality of life questionnaire that measures the functional (physical, emotional, and social) problems troublesome to adults with allergies. The RQLQ has 28 questions in 7 domains (activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms and emotional). All 28 questions were evaluated by the participant in an assessment diary over 2 weeks of treatment period and was rated on a 7-point severity scale ranging from 0 to 6, where 0=least severe to 6=extremely severe. Overall mean was calculated by summing all 28-item scores and dividing by total number of items in the questionnaire. RQLQ score ranges from 0-6 with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms. Baseline was defined as the value on Day 1 pre- dose. Change from baseline was calculated by subtracting baseline (Day 1 pre-dose) values from individual post-randomization values. Adjusted mean is reported as LS mean.
Time Frame: Baseline (Day 1 pre-dose) and Day 14 of each period
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Groups:
- Placebo: Participants received repeat doses of matching placebo once daily for 14 days in each of the 2 treatment periods, where participants were randomized to any of the two treatment sequences (active/placebo or placebo/active) separated by at least 4 weeks of washout period.
- SB-705498 12 mg: Participants received repeat doses of intranasal spray of SB-705498 12 mg as an active intervention once daily for 14 days in each of the 2 treatment periods, where participants were randomized to any of the two treatment sequences (active/placebo or placebo/active) separated by at least 4 weeks of washout period.
Arm/Group | Placebo | SB-705498 12 mg
Number analyzed (Participants) | 38 | 38
Scores on scale | -0.15 (0.126) | -0.20 (0.126)
Statistical Analysis 1: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for Day 14 in AR; Test type: Superiority or Other; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.36 to 0.26], Standard Error of Mean 0.15

10. Secondary Outcome: Mean Total Ocular Symptom Score (TOSS; Red, Itchy and Tearing Eyes) Elicited by a 1 h CDA Challenge at 1 h Post-dose on Day 1, 1 and 24 h Post-dose on Day 14 to Compare the Effect of Intranasal SB-705498 12 mg Compared With Placebo
Description: The assessment of TOSS was done based on a CDA challenge, for 1 h in a controlled environmental exposure chamber which was validated for 14+/-5 degree C, <15% relative humidity and 5+/-3 ft/sec air velocity, 1 h post dose on Day 1 and 1 h and 24 h post dose on Day 14 (Day 15). TOSS was calculated as the sum of the symptom scores for 3 ocular symptoms of itching/burning eyes, tearing/watering eyes, and redness of eyes. It was rated on a 4-point severity scale ranging from 0 to 3, where: 0=absent, 1=mild, 2=moderate and 3=severe (symptom hard to tolerate, interferes with daily activities/sleeping). TOSS score ranges from 0-9 with 0 representing an absence of symptoms and 9 representing severe symptoms. These values were used to derive the WM (s) of the CDA challenge value and the maximum score. WM is reported as LS mean.
Time Frame: Day 1 and 15 of each period (Day 14, 24 h post- dose was assessed on Day 15)
Population: All Subjects Population. Only those participants available at the specified time points was analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Placebo | SB-705498 12 mg
Number analyzed (Participants) | 38 | 40
Scores on scale
  WM 0-60 TOSS, Day 1 | 1.99 (0.273) | 2.26 (0.272)
  WM 0-60 TOSS, Day 14, 1 h: number analyzed (Participants) | 37 | 39
  WM 0-60 TOSS, Day 14, 1 h | 2.05 (0.276) | 2.16 (0.272)
  WM 0-60 TOSS, Day 14, 24 h: number analyzed (Participants) | 38 | 38
  WM 0-60 TOSS, Day 14, 24 h | 1.91 (0.261) | 2.12 (0.261)
  Maximum TOSS, Day 1, 1 h | 3.08 (0.366) | 3.27 (0.364)
  Maximum TOSS, Day 14, 1 h: number analyzed (Participants) | 37 | 39
  Maximum TOSS, Day 14, 1 h | 2.81 (0.350) | 3.07 (0.344)
  Maximum TOSS, Day 14, 24 h: number analyzed (Participants) | 38 | 38
  Maximum TOSS, Day 14, 24 h | 2.86 (0.355) | 3.15 (0.354)
Statistical Analysis 1: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for Day 1, 1 h in WM 0-60 TOSS; Test type: Superiority or Other; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.06 to 0.60], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for Day 14, 1 h in WM 0-60 TOSS; Test type: Superiority or Other; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.32 to 0.53], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for Day 14, 24 h in WM 0-60 TOSS; Test type: Superiority or Other; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.22 to 0.63], Standard Error of Mean 0.21
Statistical Analysis 4: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for Day 1, 1 h in Maximum TOSS; Test type: Superiority or Other; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.30 to 0.68], Standard Error of Mean 0.24
Statistical Analysis 5: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for Day 14, 1 h in Maximum TOSS; Test type: Superiority or Other; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-0.34 to 0.86], Standard Error of Mean 0.30
Statistical Analysis 6: Comparison: Placebo vs SB-705498 12 mg; Placebo vs SB-705498 12 mg for Day 14, 24 h in Maximum TOSS; Test type: Superiority or Other; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-0.15 to 0.73], Standard Error of Mean 0.22

11. Secondary Outcome: Pharmacokinetic Parameter of Area Under the Plasma Concentration-time Curves From Time Zero (Pre- Dose) to 3 h and 24 h (t) on Day 1 and Day 14 (AUC [0-3], AUC [0-t])
Description: Blood samples for pharmacokinetic assessment were collected at pre-dose (0 h), 1, 2, 3 and 24 h post-dose on Day 1 and Day 14 of each period. The area under the plasma concentration-time curves from time zero (pre- dose) to 3 h, AUC (0-3) and the last quantifiable concentration, AUC (0-t) (24 h) was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. The AUC of non-calculable (NC) due to non-quantifiable concentration measured as below lower limit of quantification (NQ) values were imputed by 0.5 x lowest observed AUC (i.e., AUC [0-3]: 0.5 x 6.4; AUC[0-t]: 0.5 x 6.3). Coefficient of variation (CVb [%]) was calculated as, CVb (%) = SQRT (exp [SD2-1]) x 100, where SQRT is the square root, exp is the exponent and SD is the standard deviation of the logarithmically transformed data. Analysis was done on the number of participants with non-missing observations (including imputed NC values).
Time Frame: Pre-dose (0 h), 1, 2, 3 and 24 h post-dose on Day 1 and Day 14 of each period.
Population: Analysis was done on Pharmacokinetic Population, defined as participants in the 'All Subjects' population for whom a pharmacokinetic sample was obtained and analysed. Imputed NC values were derived for AUC (0-3), on Day 1 for 3 participants and for AUC (0-t) on Day 1 for 2 participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram × hour per milliliter (ng*h/mL)
Arm/Group | SB-705498 12 mg
Number analyzed (Participants) | 39
Nanogram × hour per milliliter (ng*h/mL)
  AUC (0-3), Day 1 | 64.01 (197.5)
  AUC (0-3), Day 14 | 144.46 (107.7)
  AUC (0-t), Day 1 | 65.08 (186.5)
  AUC (0-t), Day 14 | 950.47 (125.1)

12. Secondary Outcome: Pharmacokinetic Parameter of Maximum Observed Plasma Concentration (Cmax) on Day 1 and 14
Description: Blood samples for pharmacokinetic assessment were collected at pre-dose (0 h), 1, 2, 3 and 24 h post-dose on Day 1 and Day 14 of each period. The first occurrence of Cmax was determined directly from the raw concentration-time data on Day 1 and Day 14 where, NQs were imputed to zero or missing and lower limit of quantification was 2.5 nanogram per millilitre (ng /mL). Logarithmically transformed data is reported for Cmax. CVb (%) was calculated as, CVb (%) = SQRT (exp [SD2-1]) x 100, where SD is the standard deviation of the logarithmically transformed data. Analysis was done on the number of participants with non-missing observations (including imputed NC values).
Time Frame: Pre-dose (0 h), 1, 2, 3 and 24 h post-dose on Day 1 and Day 14 of each period.
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | SB-705498 12 mg
Number analyzed (Participants) | 39
ng/mL
  Day 1 | 44.040 (152.3)
  Day 14 | 72.800 (111.5)

13. Secondary Outcome: Pharmacokinetic Parameter of Time to Maximum Observed Plasma Concentration (Tmax) on Day 1 and 14
Description: Blood samples for pharmacokinetic assessment were collected at pre-dose (0 h), 1, 2, 3 and 24 h post-dose on Day 1 and Day 14 of each period. Tmax was determined directly from the raw concentration-time data on Day 1 and Day 14 where, NQs were imputed to zero or missing and lower limit of quantification is 2.5 ng /mL. Analysis was done on the number of participants with non-missing observations (including imputed NC values)
Time Frame: Pre-dose (0 h), 1, 2, 3 and 24 h post-dose on Day 1 and Day 14 of each period.
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: h
Arm/Group | SB-705498 12 mg
Number analyzed (Participants) | 39
h
  Day 1 | 2.0000 [0.983 to 3.033]
  Day 14 | 2.9833 [0.983 to 3.083]

14. Secondary Outcome: Number of Participants With Any Adverse Event (AE), Serious Adverse Event or Drug-related AE
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition, associated with liver injury and impaired liver function defined as alanine aminotransferase >=3 x upper limit of normal (ULN), and total bilirubin >=2 x ULN or international normalised ratio >1.5. AEs were classified as potentially drug-related, based on the investigator's judgement.
Time Frame: Start of study treatment (Day 1 of first period) up to follow up, for up to 28 days.
Population: All Subjects Population.
Measure: Number; unit: Participants
Groups:
- SB-705498 12 mg: Participants received repeat doses of intranasal spray of SB-705498 12 milligram (mg) as an active intervention once daily for 14 days in each of the 2 treatment periods, where participants were randomized to any of the two treatment sequences (active/placebo or placebo/active) separated by at least 4 weeks of washout period.
Arm/Group | Placebo | SB-705498 12 mg
Number analyzed (Participants) | 38 | 39
Participants
  Any AE | 8 | 9
  Any SAE | 0 | 0
  Drug- related AE | 2 | 1

15. Secondary Outcome: Number of Participants With Abnormal (Both Not Clinically Significant and Clinically Significant) Electrocardiogram (ECG) Findings
Description: ECGs were obtained on Day 1 (pre-dose) and Day 14 (pre- dose) of each period. Single 12-lead ECGs was obtained at each timepoint during the study using an ECG machine that automatically calculated the heart rate (HR) and measures PR, QRS, QT, and QTc intervals. Participants with abnormal (not clinically significant), abnormal (clinically significant) and no result were presented.
Time Frame: Day 1 (pre-dose) and Day 14 (pre-dose)
Population: All Subjects Population.
Measure: Number; unit: Participants
Arm/Group | Placebo | SB-705498 12 mg
Number analyzed (Participants) | 38 | 39
Participants
  Abnormal - Not clinically significant, Day 1 | 6 | 3
  Abnormal - Not clinically significant, Day 14 | 2 | 2
  Abnormal - Clinically significant, Day 1 | 0 | 0
  Abnormal - Clinically significant, Day 14 | 0 | 0
  No result, Day 1 | 2 | 2
  No result, Day 14 | 1 | 0

16. Secondary Outcome: Number of Participants With Haematology Abnormalities of Potential Clinical Importance (PCI) at Any Time During Treatment
Description: The PCI values of hematology parameters were obtained by multiplying a fixed factor to the site's upper or lower limit normal ranges for each of the parameter. The factors were white blood cell count (WBC): 0.67 for relative low; 1.82 for relative high, haemoglobin (Hb) relative high: male - 1.03; female - 1.13, haematocrit (relative high): male - 1.02; female - 1.17, platelets: 0.67 for relative low; 1.57 for relative high, neutrophils (relative low): 0.83, lymphocytes (relative low): 0.81.
Time Frame: Day 14 of each period
Population: All Subjects Population.
Measure: Number; unit: Participants
Arm/Group | Placebo | SB-705498 12 mg
Number analyzed (Participants) | 38 | 39
Participants
  Total neutrophils, PCI- Low | 1 | 2
  Lymphocytes, PCI- Low | 0 | 2

17. Secondary Outcome: Number of Participants With Clinical Chemistry PCI Abnormalities of Albumin, Calcium, Glucose, Potassium, Sodium and Total Carbon Dioxide (CO2) at Any Time During Treatment
Description: The PCI values of albumin, calcium, glucose, potassium, sodium and total CO2 were obtained by multiplying a fixed factor to the site's upper or lower limit normal ranges for each of the parameter. The factors were albumin (relative low): 0.86, calcium: 0.91 for relative low; 1.06 for relative high, glucose: 0.71 for relative low; 1.41 for relative high, potassium: 0.86 for relative low; 1.10 for relative high, sodium: 0.96 for relative low; 1.03 for relative high and total CO2: 0.86 for relative low; 1. 14 for relative high.
Time Frame: Day 14 of each period
Population: All Subjects Population.
Measure: Number; unit: Participants
Arm/Group | Placebo | SB-705498 12 mg
Number analyzed (Participants) | 38 | 39
Participants | 0 | 1

18. Secondary Outcome: Number of Participants With Clinical Chemistry PCI Abnormalities of Creatinine, Blood Urea Nitrogen (BUN), Uric Acid, Cholesterol, Triglycerides, Lactate Dehydrogenase (LDH) and Liver Function Test at Any Time During Treatment
Description: The PCI values of clinical chemistry parameters were creatinine: low- male is <75 micromoles per litre (mcmol/L); low- female is <65 mcmol/L; high- male >110 mcmol/L; high- female >95 mcmol/L, BUN: high is >1.5 x ULN millimole per litre (mmol/L), uric acid: low- male is <180 mcmol/L; low- female is <120 mcmol/L; high- male >480 mcmol/L; high- female >420 mcmol/L, cholesterol: low is <3.9 mmol/L; high is >6.5 mmol/L [if age <=40, if age >40- high is >6.55 mmol/L], triglycerides: low- <0.5 mmol/L; high- >2.0 mmol/L, LDH: >220 units per lire (U/L). For high alanine aminotransferase (ALT); aspartate aminotransferase (AST); alkaline phosphatase is >=2 x ULN U/L. Total bilirubin high is >=1.5 x ULN mcmol/L, gamma glutamyltransferase (GGT) high: male- >60 U/L; female > 40 U/L.
Time Frame: Day 14 of each period
Population: All Subjects Population.
Measure: Number; unit: Participants
Arm/Group | Placebo | SB-705498 12 mg
Number analyzed (Participants) | 38 | 39
Participants
  Creatinine, High | 1 | 0
  Uric acid, High | 1 | 0
  GGT, High | 2 | 2

19. Secondary Outcome: Number of Participants With Vital Sign of Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP), HR and Body Temperature of PCI Abnormalities at Any Time During Treatment
Description: The PCI values of vital signs were SBP: <85 and >160 millimetres of mercury (mmHg), DBP of <45 and >100 mmHg, HR of <40 and >110 beats per minute (bpm) and body temperature of <36 and >37.5oC.
Time Frame: Day 1 and Day 14 of each period
Population: All Subjects Population.
Measure: Number; unit: Participants
Arm/Group | Placebo | SB-705498 12 mg
Number analyzed (Participants) | 38 | 39
Participants
  SBP, Low | 0 | 1
  HR, High | 1 | 2
  Body temperature, Low | 7 | 14

ADVERSE EVENTS:
Time Frame: AE(s) were collected from start of study treatment (Day 1 of first period) up to follow up (up to 28 days)
Description: All Subjects population
Arm/Group | Placebo | SB-705498 12 mg
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/39
Other Adverse Events (participants affected / at risk) | 8/38 | 9/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=38) | SB-705498 12 mg (N=39)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Tonsillitis (Infections and infestations) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.